CLINICAL TRIAL: NCT00004917
Title: A Randomized Phase III Trial to Assess the Effect of Erythropoietin on Local-Regional Control in Anemic Patients Treated With Radiotherapy for Carcinoma of the Head and Neck
Brief Title: Radiation Therapy With or Without Epoetin Alfa in Treating Anemic Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RTOG-9903; CDR0000067599
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2016-12

CONDITIONS: Anemia; Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; anemia
MeSH Terms: conditions — Anemia; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Epoetin Alfa; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: epoetin alfa
Drug: cisplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Epoetin alfa may stimulate red blood cell production and treat anemia in patients with head and neck cancer. It is not yet known whether receiving radiation therapy with epoetin alfa is more effective than radiation therapy alone in treating anemic patients with head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without epoetin alfa in treating anemic patients who have head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether epoetin alfa given during definitive radiotherapy or chemoradiotherapy improves the local-regional control rate in anemic patients with squamous cell carcinoma of the head and neck.

Secondary

* Determine whether this drug improves survival in this patient population.
* Identify patterns in first failure in these patients.
* Determine whether there is a significant increase in hemoglobin level between the baseline value and the value at 28 days after starting epoetin alfa in these patients.
* Assess the toxicity of this regimen in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to stage (I/II vs III/IV without chemotherapy vs III/IV with chemotherapy), pretreatment hemoglobin level (9.0 to less than 11.5 g/dL vs 11.5 to 13.5 g/dL), and gender. Patients are randomized to one of two treatment arms.

* Arm I: Patients with stage I or II disease undergo radiotherapy once daily for 6-7 weeks. Patients with stage III or IV disease undergo radiotherapy once daily for 3.5 weeks and then twice daily (6 hours apart) for 2.5 weeks for a total of 6 weeks.
* Arm II: Patients undergo radiotherapy as in arm I. Beginning 7-10 days before radiotherapy, patients receive epoetin alfa subcutaneously once weekly until the end of radiotherapy.

Patients with stage III/IV disease may receive concurrent cisplatin IV over 1-2 hours on days 1 and 22 of radiotherapy.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 372 patients (186 per arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive squamous cell carcinoma of the head and neck, including carcinoma arising from the oral cavity, oropharynx, larynx, and hypopharynx

  * Stage I-IV disease
  * No distant metastases
  * No carcinoma of the nasopharynx, nasal cavity/paranasal sinuses, or salivary glands
  * No carcinoma in situ without an identifiable invasive component
* Plan for radiotherapy in continuous course
* Prior surgical exploration with gross residual disease remaining allowed
* Prior neck dissection with or without biopsy of primary tumor, but no radical surgery for primary tumor, allowed
* Anemia, defined as hemoglobin no greater than 13.5 g/dL for males and no greater than 12.5 g/dL for females (transfusion prior to study allowed)

  * No severe anemia (i.e., hemoglobin less than 9.0 g/dL)
  * No anemia confirmed to be due to causes other than chronic disease (e.g., iron deficiency anemia)
* Not entered on other RTOG head and neck protocols

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Stage III/IV patients receiving concurrent cisplatin:

  * Absolute neutrophil count at least 2,000/mm^3
  * Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Stage III/IV patients receiving concurrent cisplatin:

  * Creatinine no greater than 1.5 mg/dL
  * Creatinine clearance at least 50 mL/min

Cardiovascular:

* No malignant or poorly controlled hypertension (e.g., symptomatic hypertension or diastolic blood pressure of 100 mm Hg or greater despite antihypertensive medication)
* No unstable angina or other poorly controlled cardiac disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* If stage III or IV disease is present, willing to come for twice daily radiotherapy for the last 2.5 weeks of therapy
* No active infection requiring IV antibiotics
* No unexplained fever
* No AIDS or other history of congenital or acquired immunodeficiency
* No other malignancies within the past 3 years except carcinoma in situ or nonmelanomatous skin cancer
* No known hypersensitivity to mammalian cell-derived products or to human albumin
* No acute/subacute illness that would make the need for transfusion likely

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since other prior cytokine therapy (e.g., filgrastim [G-CSF], interleukins, or interferons)
* No prior epoetin alfa
* No other concurrent cytokine therapy

Chemotherapy:

* No prior chemotherapy
* Concurrent cisplatin, paclitaxel/cisplatin, or paclitaxel/carboplatin for patients with stage III/IV disease is allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to the head and neck

Surgery:

* See Disease Characteristics

Other:

* No concurrent amifostine
* No concurrent transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2007-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Machtay, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (261):
- United States (240):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Robert and Beverly Lewis Family Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Incorporated, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Torrance Memorial Medical Center, Torrance, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Florida Radiation Oncology Group, Jacksonville, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - CCOP - Scott and White Hospital, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarian Health Partners Inc., Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Cancer Center at Lexington Clinic, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - NSMC Cancer Center, Peabody, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Fairview University Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center - Omaha, Omaha, Nebraska
  - Nebraska Health System, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Medical Center of Princeton, Princeton, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Cancer Center, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Arlington Cancer Center, Arlington, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Jin Soo Lee Practice Inc., Gyeonggi-do, South Korea

REFERENCES:
- [Result] Machtay M, Pajak TF, Suntharalingam M, Shenouda G, Hershock D, Stripp DC, Cmelak AJ, Schulsinger A, Fu KK; Radiation Therapy Oncology Group. Radiotherapy with or without erythropoietin for anemic patients with head and neck cancer: a randomized trial of the Radiation Therapy Oncology Group (RTOG 99-03). Int J Radiat Oncol Biol Phys. 2007 Nov 15;69(4):1008-17. doi: 10.1016/j.ijrobp.2007.04.063. Epub 2007 Aug 23. PMID 17716826
- [Result] Machtay M, Pajak T, Suntharalingam M, et al.: Definitive radiotherapy +/- erythropoietin for squamous cell carcinoma of the head and neck: preliminary report of RTOG 99-03. [Abstract] Int J Radiat Oncol Biol Phys 60 (Suppl 1): A-5, S132, 2004.